CLINICAL TRIAL: NCT00347464
Title: Adaptive Behavior Assessment of Men With 49, XXXXY, Klinefelter Syndrome
Status: Withdrawn | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 2005-295
Record Dates: First submitted 2006-06-29; First posted 2006-07-04 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Klinefelter Syndrome
Keywords: Kleinfelter
MeSH Terms: conditions — Klinefelter Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Klinefelter syndrome, a congenital chromosomal abnormality with one or more extra X chromosomes, occurs in out of 400 live male births. The majority of Klinefelter men present with a 47, XXY karyotype. The "poly-X variant", with the 49,XXXXY karyotype is uncommon. This syndrome, where subjects have two or more X chromosomes presents with primary hypogonadism, and, particularly if associated with the 49,XXXXY karyotype, significantly impacts life skills across a variety of dimensions, including areas of communication, community use, functional academics, home/school living, health and safety, leisure, self-care, self direction, and work. Adaptive behavior abnormalities in 46,XXY men are well known and described. In the poly-X variant of the 49,XXXXY karyotype, adaptive behavior abnormalities are expected to be much more significant, making these patients eligible for services and Social Security benefits.

In 49,XXXXY men no study to date has examined these areas of inquiry in a large patient population, using a psychometrically sound instrument in a large patient population. Current publications are limited to individual case reports or small case summaries. It is important to study the adaptive behavior in its highly abnormal presentation in 49,XXXXY men in order to learn more about the effect of additional X chromosomes on adaptive skills, which determine how an individual responds to daily demands and in order to develop treatment and training goals.

ELIGIBILITY:
Inclusion Criteria:

* Any Klinefelter male with proven 49,XXXXY karyotype, who does not present with and is not being treated for significant physical/mental illness which might affect his adaptive behavior, who or whose parent or primary caretaker is able to provide informed consent to participate in the study and who or whose parent or primary caretaker has adequate command of the English language, to provide meaningful information will be invited to participate in this study.

Ages: 2 Years to 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Klinefelter males ages 2-21 with proven 49,XXXXY karyotype
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-06; Study Completion 2008-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfram E Nolten, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States